CLINICAL TRIAL: NCT04345874
Title: Compliance and Technical Assistance for Child and Adult Care Food Program in Family Child Care Homes- Virtual Implementation
Brief Title: Virtual Technical Assistance for Child and Adult Care Food Program in Family Child Care Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10747
Record Dates: First submitted 2020-04-06; First posted 2020-04-15 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Nutrition Poor; Health Behavior
Keywords: early childhood education; family childcare home; food environment
MeSH Terms: conditions — Malnutrition; Health Behavior

STUDY DESIGN:
Intervention Model Description: Randomized trial where family child care home providers are randomized to either nutrition or environmental health technical assistance intervention. Interventions are matched for time and contact.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrition technical assistance (Experimental): three encounters with Intervention team over three months: two virtual 60-90 minutes visits one-on-one with the FCCH each scheduled at the convenience of the provider and a 3- hour virtual group class with other providers.
  Interventions: Behavioral: Nutrition technical assistance
- Children's environmental health technical assistance (Experimental): three encounters with Intervention team over three months: two virtual 60-90 minutes visits one-on-one with the FCCH each scheduled at the convenience of the provider and a 3- hour virtual group class with other providers.
  Interventions: Behavioral: Children's environmental health technical assistance

INTERVENTIONS:
Behavioral: Nutrition technical assistance — Participating family child care home providers in rural counties will be randomized to either the Nutrition Intervention (n=27), or an environmental health comparison group (n=27) that will receive an Integrated Pest Management and Green Cleaning intervention with the same format and visit frequency. Briefly, the Nutrition Technical Assistance Intervention and comparison group will consist of three encounters with our intervention team: two 60-90 minutes virtual one-on-one visits scheduled at the convenience of the family child care home provider and a 3-hour virtual group class session with other providers. Total contact time with intervention staff will be 6 hours. All participants will receive a toolkit. Providers will complete either intervention virtually over a period of three months.
  Arms: Nutrition technical assistance
Behavioral: Children's environmental health technical assistance — Participating family child care home providers in rural counties will be randomized to either the Nutrition Intervention (n=27), or an environmental health comparison group (n=27) that will receive an Integrated Pest Management and Green Cleaning intervention with the same format and visit frequency. Briefly, the Nutrition Technical Assistance Intervention and comparison group will consist of three encounters with our intervention team: two 60-90 minutes virtual one-on-one visits scheduled at the convenience of the family child care home provider and a 3-hour virtual group class session with other providers. Total contact time with intervention staff will be 6 hours. All participants will receive a toolkit. Providers will complete either intervention virtually over a period of three months.
  Arms: Children's environmental health technical assistance

SUMMARY:
This study evaluates the effect of a fully virtual nutrition technical assistance training program for family child care home providers on the food they serve young children in their care and the food environment in their home. Half the providers will be randomly assigned to the nutrition program and the other half will receive a comparison on environmental health.

DETAILED DESCRIPTION:
Early care and education (ECE) providers play a vital role in ensuring that young children have access to nutritious foods. Over 25% of children in ECE (1.2 million children) attend Family Child Care Homes (FCCH). Improvements in the Child and Adult Care Food Program (CACFP) may introduce new barriers for FCCH, which have limited meal preparation capacity. Limited research has examined foods served by FCCH providers, and no group randomized trials have been conducted using a Community-Based Participatory approach in FCCH and including an evaluation of intervention costs.

Goals: 1. Determine the effectiveness of a virtual, rural outreach community-based Nutrition Technical Assistance Intervention to enhance meeting CACFP best-practices.

Methods: Conduct a cross-sectional assessment of a random sample of FCCH providers' (n=54) menus and meals served. Foods will be evaluated against the CACFP requirements and best-practices. Trained Extension Educators will implement both interventions (n=27 intervention, n=27 comparison) focused in rural counties, reaching underserved rural and low-income populations. The intervention is based on theoretical foundations and formative interviews, and will consist of two virtual 60-90-minute one-on-one visits with the FCCH and one virtual group class lasting approximately 3 hours.

ELIGIBILITY:
Inclusion Criteria:

* Family Child Care Home Providers who participate in the Child and Adult Care Food Program in Oklahoma.
* Providers must serve at least 1 2-to-5 year old child and speak English.
* Providers must plan to continue their business while participating in CACFP for the next 12 months.

Exclusion Criteria:

* Family Child Care Home Providers who care for only infants and toddlers and not speak English.
* Participant withdraws.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2021-12-07 (Actual)

PRIMARY OUTCOMES:
Self-reported nutrition practices | baseline, changes post 3-months, changes post 12-months
  Providers report the frequency and type of fruit and vegetables, milk, and salty snacks served using the NAPSACC Self-Report tool virtually/on-paper, tailored for FCCH
nutrition environment | baseline, changes post 3-months, changes post 12-months
  Self-reporting the EPAO survey virtually/on-paper
compliance of menu and meal with Child and Adult Care Food Program requirements using compliance scoring tool created by collaborative research team | baseline, changes post 3-months, changes post 12-months
  menus and meals served are compared to the requirements and best practices of the CACFP using compliance scoring tool created by the collaborative research team
dietary quality of foods served | baseline, changes post 3-months, changes post 12-months
  analysis of remote food photograph of a child's breakfast, lunch, snack

SECONDARY OUTCOMES:
Provider self-efficacy | baseline, post 3-months, post 12-months
  providers will self report nutrition and environmental health self-efficacy using using survey created by the collaborative research team virtually/on-paper
Environmental health observation | baseline, post 3-months, post 12-months
  observation of household cleaners and chemicals and signs of pests virtually, a tool created by the collaborative research team

CONTACTS AND LOCATIONS:
Overall Officials: Susan B Sisson, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States